CLINICAL TRIAL: NCT01222234
Title: Impact of Vitamin D Therapies on Monocyte Function in Chronic Kidney Disease
Brief Title: Impact of Vitamin D Therapies on Chronic Kidney Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Kansas Medical Center (Other)
Responsible Party: Principal Investigator, Jason Stubbs, MD, Assistant Professor, University of Kansas Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 11936
Record Dates: First submitted 2010-10-13; First posted 2010-10-18 (Estimated); Results first posted 2016-05-16 (Estimated); Last update posted 2016-05-16 (Estimated); Status verified 2016-04

CONDITIONS: Chronic Kidney Disease (CKD); End-stage Renal Disease (ESRD)
MeSH Terms: conditions — Renal Insufficiency, Chronic; Kidney Failure, Chronic | interventions — Cholecalciferol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Group 1: Cholecalciferol - CKD (Experimental): Patients in this group have low vitamin D levels and Chronic Kidney Disease (CKD). They will be administered cholecalciferol 50,000 IU twice weekly for 8 weeks.
  Interventions: Drug: Cholecalciferol - CKD
- Group 2: Calcitriol - CKD (Experimental): Patients in this group have low vitamin D levels and Chronic Kidney Disease (CKD). They will be administered calcitriol 0.25mcg daily for 8 weeks.
  Interventions: Device: Calcitriol - CKD
- Group 3: Cholecalciferol - non-CKD (Experimental): Patients in this arm have low vitamin D levels and normal kidney function. They will be administered cholecalciferol 50,000 IU twice weekly for 8 weeks.
  Interventions: Drug: Cholecalciferol - non-CKD

INTERVENTIONS:
Drug: Cholecalciferol - CKD — Cholecalciferol tablet 50,000 IU twice weekly for 8 weeks
  Other Names: Vitamin D3
  Arms: Group 1: Cholecalciferol - CKD
Device: Calcitriol - CKD — Calcitriol 0.25 mcg once daily for 8 weeks
  Other Names: 1,25(OH)2D
  Arms: Group 2: Calcitriol - CKD
Drug: Cholecalciferol - non-CKD — Cholecalciferol tablet 50,000 IU twice weekly for 8 weeks
  Other Names: Vitamin D3
  Arms: Group 3: Cholecalciferol - non-CKD

SUMMARY:
This investigation will consist of a prospective study utilizing two separate populations of patients with 25(OH)D deficiency, one population with chronic kidney disease (CKD) and one with normal renal function.

DETAILED DESCRIPTION:
Vitamin D helps form and strengthens bones by allowing the body to absorb calcium. Vitamin D helps the immune system fight infection as well as helps keep muscles strong. Without enough vitamin D, bones can become weak, thin and brittle.

Vitamin D is useful in people with all different types of health issues. CKD is the slow loss of kidney function over time. The main function of the kidneys is to remove wastes and excess water from the body. This loss of function usually takes months or years to occur Patients with CKD often have low levels of vitamin D in their blood.

This study will have two groups of patients with CKD and one group of patients that have normal kidney function, but all groups will have low levels of vitamin D. The two groups with CKD (group 1 and group 2) will receive either cholecalciferol or calcitriol. The purpose of having a control group (group 3) without CKD will be to evaluate if any changes that are witnessed in response to vitamin D therapy are specific to patients with kidney disease or apply to all patients with vitamin D deficiency who receive vitamin D supplements.

There are two different drugs in this study. One is called Calcitriol and is approved by the Food and Drug Administration (FDA) as a vitamin D supplement. The other drug is called cholecalciferol and it is approved by the FDA. Unlike calcitriol, cholecalciferol is a nutritional form of vitamin D that can often be found in various types of foods and its chemical structure must be changed by the body to become the active form of vitamin D. It is believed that cholecalciferol may have different effects in the body compared to calcitriol. It is possible that CKD patients would benefit from receiving both of these drugs, but this is currently unclear. While on this study you will receive either one of these study drugs, depending on which group you are assigned to.

ELIGIBILITY:
Inclusion Criteria:

* Chronic kidney disease w/GFR<35ml/min
* Nutritional vitamin D deficiency, defined as 25(OH)D < 25ng/ml
* Secondary hyperparathyroidism, PTH>75pg/mL

Exclusion Criteria:

* Active infection
* Recent hospitalization for acute illness (within last month)
* Refusal to study participation
* History of chronic inflammatory disease process (i.e. inflammatory bowel, rheumatoid arthritis, SLE, etc.)
* Allergy to cholecalciferol or calcitriol
* History of parathyroidectomy
* Functional renal transplant within 5 years
* Current treatment with immunosuppressant medications
* Noncompliance with prescribed medications

Ages: 21 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2010-10; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jason Stubbs, MD, Principal Investigator — University of Kansas Medical Center
Locations (1):
- University Of Kansas Medical Center, Kansas City, Kansas, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Group 1: Cholecalciferol: Patients in this group have low vitamin D levels and Chronic Kidney Disease (CKD). Patients will be randomized to group 1 or group 2.
  Cholecalciferol: Cholecalciferol tablet, 50,000 units twice a week
- Group 2: Calcitriol: Patients in this group have low vitamin D levels and Chronic Kidney Disease (CKD). Patients will be randomized to group 1 or group 2.
  calcitriol: calcitriol 0.25 mcg every day
- Group 3: Cholecalciferol: Patients in this arm have low vitamin D levels and normal kidney function. They will be put into group 3.
  Cholecalciferol: Cholecalciferol tablet, 50,000 units twice a week
Period: Overall Study
Arm/Group | Group 1: Cholecalciferol | Group 2: Calcitriol | Group 3: Cholecalciferol
Started | 15 | 17 | 24
Completed | 15 | 15 | 22
Not Completed | 0 | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1: Cholecalciferol | Group 2: Calcitriol | Group 3: Cholecalciferol | Total
Number analyzed (Participants) | 15 | 17 | 24 | 56
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 9 | 11 | 20 | 40
  >=65 years | 6 | 6 | 4 | 16
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.1 (13.3) | 59.8 (11.6) | 48.5 (14.2) | 56.1 (13.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 10 | 21 | 40
  Male | 6 | 7 | 3 | 16
Region of Enrollment [Number; unit: participants]
  United States | 15 | 17 | 24 | 56

OUTCOME MEASURES:

1. Primary Outcome: Monocyte Protein Expression
Description: Flow cytometry analysis of monocyte CD14, ACE, VDR, and Mac-1 expression
Time Frame: 8 weeks of therapy
Population: The primary comparison for this outcome was between only CKD groups (groups 1 and 2); therefore data from the non-CKD group (group 3) was not analyzed for this outcome. Only 15 patients per group had data analyzed for this outcome of interest; thus, the number analyzed per group differs from the enrolled numbers.
Measure: Mean (Standard Deviation); unit: relative fluorescence units
Groups:
- Group 1: Cholecalciferol - CKD: Patients in this group have low vitamin D levels and Chronic Kidney Disease (CKD). Patients will be randomized to group 1 or group 2.
  Cholecalciferol 50,000 IU twice weekly for 8 weeks
- Group 2: Calcitriol - CKD: Patients in this group have low vitamin D levels and Chronic Kidney Disease (CKD). Patients will be randomized to group 1 or group 2.
  Calcitriol 0.25 mcg every day
Arm/Group | Group 1: Cholecalciferol - CKD | Group 2: Calcitriol - CKD
Number analyzed (Participants) | 15 | 15
relative fluorescence units
  CD14 | 34110 (9372) | 38540 (16880)
  ACE | 1359 (347.2) | 1360 (290.8)
  VDR | 2799 (1210) | 3468 (3123)
  Mac-1 | 14318 (4196.4) | 14278.5 (4891.3)

2. Primary Outcome: Change in 24,25(OH)2D Levels in CKD vs. Non-CKD Subjects Receiving Cholecalciferol
Time Frame: 8 weeks of therapy
Population: The primary comparison for this outcome of interest was between subjects taking cholecalciferol, so the calcitriol group (group 2) was excluded from the analysis. Only 15 patients per group had data analyzed for this outcome of interest; thus, the number analyzed per group differs from the enrolled numbers.
Measure: Mean (Standard Deviation); unit: ng/ml
Groups:
- Group 1: CKD Cholecalciferol: Patients in this group have low vitamin D levels and Chronic Kidney Disease (CKD). Patients will be randomized to group 1 or group 2.
  Cholecalciferol: Cholecalciferol tablet, 50,000 units twice a week
- Group 3: Non-CKD Cholecalciferol: Patients in this arm have low vitamin D levels and normal kidney function. They will be put into group 3.
  Cholecalciferol: Cholecalciferol tablet, 50,000 units twice a week
Arm/Group | Group 1: CKD Cholecalciferol | Group 3: Non-CKD Cholecalciferol
Number analyzed (Participants) | 15 | 15
ng/ml | 1.59 (0.73) | 3.59 (1.14)

ADVERSE EVENTS:
Arm/Group | Group 1: Cholecalciferol | Group 2: Calcitriol | Group 3: Cholecalciferol
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/17 | 0/24
Other Adverse Events (participants affected / at risk) | 0/15 | 1/17 | 1/24
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1: Cholecalciferol (N=15) | Group 2: Calcitriol (N=17) | Group 3: Cholecalciferol (N=24)
constipation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
diarrhea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes